CLINICAL TRIAL: NCT05501626
Title: Evaluation of Theta-burst Stimulation Efficacy, Safety and Tolerability in Major Depressive Episodes of Bipolar I Disorder: Randomized, Controlled, Double-blind, Parallel-group Clinical Trial
Brief Title: Evaluation of Theta-burst Stimulation Efficacy, Safety and Tolerability in Major Depressive Episodes of Bipolar I Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Ricardo Alberto Moreno, M.D., Ph.D., Professor Ricardo Moreno, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: StudyTBS
Record Dates: First submitted 2022-08-11; First posted 2022-08-15 (Actual); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: Bipolar Disorder, Type 1
Keywords: randomized clinical trial; transcranial magnetic stimulation; bipolar affective disorder; major depression
MeSH Terms: conditions — Bipolar Disorder; Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active TBS arm (Active Comparator): Patients randomized to this arm will receive active TBS 5 consecutive days of the week (Monday to Friday) in the first 3 weeks and then 2 alternate days of the week (with interval of at least 1 day between sessions) for another 3 weeks comprising 21 sections.
  Interventions: Device: Active Theta Burst Stimulation (TBS)
- Sham TBS arm (Sham Comparator): Patients randomized to this arm will receive sham TBS 5 consecutive days of the week (Monday to Friday) in the first 3 weeks and then 2 alternate days of the week (with interval of at least 1 day between sessions) for another 3 weeks comprising 21 sections.
  Interventions: Device: Sham Theta Burst Stimulation (TBS)

INTERVENTIONS:
Device: Active Theta Burst Stimulation (TBS) — Each session will be comprised of ACTIVE TBS: intermittent excitatory stimulation (iTBS) in the left dorsolateral prefrontal cortex totaling 37,800 pulses.
  Arms: Active TBS arm
Device: Sham Theta Burst Stimulation (TBS) — Each session will be comprised of SHAM TBS: intermittent excitatory stimulation (iTBS) in the left dorsolateral prefrontal cortex totaling 37,800 pulses.
  Arms: Sham TBS arm

SUMMARY:
INTRODUCTION: Pharmacological treatment of major depressive episodes in bipolar disorder (BD) is characterized by suboptimal efficacy rates, poor tolerability and adherence, delayed onset of action, and iatrogenic mood swings. The use of repetitive transcranial magnetic stimulation (rTMS) has been presented as an effective, safe and well-tolerated alternative to the treatment of uni- and bipolar depressive episodes. Recently, a new rTMS protocol was introduced, theta-burst stimulation (TBS), whose studies have shown similar efficacy with a shorter time interval than conventional rTMS. Most clinical trials performed to date evaluate the use of TBS in patients with unipolar depression or mixed samples of uni and bipolar patients. The effectiveness of TBS exclusively in BD has not been properly studied. METHODS: We will perform a 6-week, double-blind, randomized, parallel-group, sham-controlled clinical trial of active or sham TBS. We will recruit 60 patients aged between 18 and 65 years with a diagnosis of BD type I in a current moderate or severe major depressive episode resistant to at least two first- or second-line pharmacological treatments, according to CANMAT guidelines. The primary outcome measure will be the assessment of TBS efficacy through difference in scores on 17-item Hamilton Depression Scale (HAM-D) from baseline until the end of week 6 of intervention between active and sham groups. KEYWORDS: randomized clinical trial; transcranial magnetic stimulation; bipolar affective disorder; major depression.

ELIGIBILITY:
Inclusion Criteria:

* Current moderate or severe major depressive episode in bipolar I disorder assessed with Hamilton Depression Rating Scale (HAM-D) score ≥ 17 points.
* Any appropriate first or second line pharmacological regimen in accordance with Canmat guidelines to treat a major depressive episode in bipolar I disorder:

Quetiapine 300 - 600 mg/dia; Lithium serum levels 0,6 - 1,2 meq/L; Lamotrigine 100 - 200 mg/dia; Lurasidone 20 - 120 mg/dia; Divalproex; Lithium/Divalproex + Lurasidone; Lithium/Divalproex + Lamotrigine; Olanzapine 5 - 20 mg/day + Fluoxetine 20 - 60 mg/day; Lithium/Divalproex + SSRI/Bupropion.

Exclusion Criteria:

* Concomitant diagnosis of other neuropsychiatric disorders such as: schizophrenia, dementias, mental retardation, organic mental disorder, or epilepsy;
* Acute suicide ideation (assessed by interview and clinical evaluation);
* Acute psychotic depression (assessed by interview and clinical evaluation);
* Suspected or confirmed pregnancy;
* Women in breastfeeding;
* Severe or unstable clinical disease;
* Previous rTMS treatment;
* Specific contraindications to TBS: previous epileptic seizures; change in electroencephalogram at some point in life; previous stroke; previous severe traumatic brain injury (with neurosurgery); metallic object on head (except mouth) as projectile piece, surgical clip, welding fragments; any implanted device (cardiac pacemaker, intravenous catheter).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-07-10 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome Measure | From baseline to week 6
  Change in Hamilton Depression Rating Scale (HAM-D)

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Psychiatry, University of Sao Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No